CLINICAL TRIAL: NCT04953819
Title: Coronary RevascUlarization in Patients With End-stage Renal dIsease on dialysiS in China: a Nationwide and multicEnter Cohort Study.
Brief Title: Coronary Revascularization in Patients With Dialysis in China
Acronym: CRUISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Department of Cardiology, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: 2020-112-K71
Record Dates: First submitted 2021-06-16; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease; Dialysis; Intervention
Keywords: dialysis; coronary artery disease; revascularization; optimal medical therapy; prognosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Catheterization; Nutrition Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Revascularization group: This group includes patients with dialysis who have received revascularization by percutaneous coronary intervention or coronary artery bypass grafting for coronary artery disease.
  Interventions: Other: Revascularization
- Medical treatment group: This group includes patients who have received medical therapy for coronary artery disease, not percutaneous coronary intervention or coronary artery bypass grafting.
  Interventions: Other: Medical therapy

INTERVENTIONS:
Other: Revascularization — Percutaneous coronary intervention and/or coronary bypass grafting for coronary artery disease
  Other Names: Catheterization or coronary bypass grafting
  Groups: Revascularization group
Other: Medical therapy — Optimal medical therapy for coronary artery disease
  Groups: Medical treatment group

SUMMARY:
China patients in end stage renal disease receiving maintenance dialysis have a high risk of cardiovascular disease (CVD), with a prevalence of 45.5% approximately, and coronary artery disease (CAD) has been identified as the most common one. It remains unclear that what their treatment status is and whether this group of patients can benefit from revascularization in China. The investigators plan to recruit around 30 hospitals from 7 regions as study centers, which represent different levels of economic development in Mainland China. The detailed information includes demographics, medical history, coronary angiogram, in-hospital treatment and procedures, short-term and long-term outcomes. The aim of the study is to provide the real world knowledge about current status of coronary revascularization and prognosis in patients with CAD and dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above and 85 or below.
* Receives peritoneal dialysis or hemodialysis more than 1-time weekly and for more than 3 months.
* Diagnosed with coronary artery disease, including STEMI, NST-ACD, stable coronary artery disease.

Exclusion Criteria:

* Pregnancy or lactation.
* Can't be cooperative because of a mental illness or other reasons.
* Malignant tumor or severe hepatic disease.
* Life expectancy is less than 1 year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study will be selected from around 30 different hospitals in 7 different areas in China.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all-cause death | the duration of hospital stay, an expected average of 2 weeks
  All-cause deaths includes cardiac death, vascular death and non-cardiovascular death.
  1. Cardiac death: any death due to proximate cardiac cause (eg, MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
  2. Vascular death: caused by noncoronary vascular causes, such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular diseases.
  3. Non-cardiovascular death: any death not covered by the above definitions, such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide, or trauma.
Incidence of all-cause death and non-fatal myocardial infarction | 12-month follow-up
  Non-fatal myocardial infarction is defined as elevated cardiac enzymes (troponin or myocardial band fraction of creatine kinase) above the upper reference limit with ischemic symptoms or electrocardiography findings indicative of ischemia that is not related to the index procedure.

SECONDARY OUTCOMES:
Incidence of all-cause death and non-fatal myocardial infarction | within 30 days after discharge
  Definitions of all-cause death and non-fatal myocardial infarction as mentioned above.
Incidence of all-cause death, non-fatal myocardial infarction, non-fatal stroke, repeat revascularization, cardiovascular rehospitalization. | 12-month follow-up
  1. Definitions of all-cause death and non-fatal myocardial infarction as mentioned above.
  2. Non-fatal stroke is defined as the rapid onset of a new persistent neurologic deficit attributed to an obstruction in cerebral blood flow and/or cerebral hemorrhage with no apparent non-vascular cause.
  3. Repeat revascularization is any unplanned repeat revascularization of either a target vessel or non-target vessel or CABG.
  4. Cardiovascular rehospitalization is rehospitalization due to MI, angina, heart failure, stroke, arrhythmia or conduction disturbance, sudden cardiac arrest and other cardiovascular problem.
Incidence of bleeding | 12-month follow-up
  Bleeding Academic Research Consortium (BARC) type 2 to 5 bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jingang Zheng, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided